CLINICAL TRIAL: NCT06527079
Title: Evaluation of Clinical Decision Support in Opioid Tapering
Status: Not yet recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-1193; 24-1193 (Other: COMIRB); R61DA057610 (NIH)
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Medication Abuse; Harm Reduction; Opioid Use Disorder; Opioid Prescribing; Opioid Overdose; Prevention
MeSH Terms: conditions — Substance-Related Disorders; Harm Reduction; Opioid-Related Disorders; Opiate Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual Care: Control group to enable tracking of temporal changes in prescribing. Providers will not see any alert.
- CDS Notification: Providers will see a clinical decision support tool within the electronic health record when treating a patient who may benefit from or is currently tapering opioid medications to encourage the provider to use a clinical care pathway that provides resources and decision support in tapering.
  Interventions: Other: Opioid Tapering Pathway Clinical Decision Support (CDS)

INTERVENTIONS:
Other: Opioid Tapering Pathway Clinical Decision Support (CDS) — Clinical decision support in the form of an electronic health record (EHR)-integrated, provider facing notification suggesting the provider utilize a clinical care pathway that provides resources and decision support in opioid tapering in line with CDC guidelines.
  Groups: CDS Notification

SUMMARY:
The 2022 Center for Disease Control and Prevention (CDC) clinical practice guideline for prescribing opioids for pain recommends that when tapering a patient's opioid dose, doses should be decreased at a slow rate to reduce the risk of withdrawal symptoms, overdose, and to promote tolerance of the tapering. This project will evaluate a clinical decision support (CDS) tool in the form of a clinical care pathway that gives providers information, recommendations, and educational material on strategies for opioid tapering. Primary care providers will be randomized at the clinic location to a control arm or intervention arm. The control arm will have the clinical care pathway available, but will not be reminded of the pathway when tapering a patient. The intervention arm will receive a nudge when prescribing a tapering opioid strategy to a patient to use the clinical care pathway. The rate of opioid tapering in line with CDC guidelines will be examined as well as long-term patient outcomes of opioid overdose or poisoning using existing patient health records. The study period will be approximately 18 months.

ELIGIBILITY:
Inclusion Criteria: Primary care patients being tapered from an opioid. Tapering patients:

* Have an active opioid prescription for more than 3 months and
* Prescribed more than 90 morphine milligram equivalents (MME) per day or
* Co-prescribed an opioid and benzodiazepine or
* Received a reduction in opioid dosage by more than 5% MME per day

Exclusion Criteria:

* Patients <12 and >89
* Patients with active cancer diagnosis in last 1 year
* Patients with hospice care/palliative care order
* Patients with sickle cell disease diagnosis

Ages: 12 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents and visitors to the state of Colorado who seek healthcare within the University of Colorado Health (UCHealth) primary care system receiving long-term opioid treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of encounters tapering within CDC guidelines | 18 months
  The number of encounters where a provider's actions are in line with CDC tapering guidelines divided by the total number of opioid tapering prescriptions

SECONDARY OUTCOMES:
Clinical decision support (CDS) acceptance rate | 18 months
  The number of times providers accepted the clinical decision support (CDS) tool and utilized the clinical care pathway
Subsequent opioid overdose/poisoning rates | 6 months after taper encounter
  The number of patients who had a diagnosis of opioid overdose or poisoning in the six months following an opioid tapering prescription
Health care utilization | 6 months after taper encounter
  The number of emergency department and clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hoppe, DO, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: Yes
De-identified data utilized in this project will be housed on the National Addiction and HIV Data Archive Program (NAHDAP) repository after final study results have been published.
Supporting Information: Study Protocol
Time Frame: Data will be provided to NAHDAP after study results are published in peer-reviewed journals.
Access Criteria: Prior to downloading study data, the individual will have to register with the site and agree to a standard data use agreement.
URL: https://www.icpsr.umich.edu/web/pages/NAHDAP/